CLINICAL TRIAL: NCT03889821
Title: Does Mindfulness Training Enhance Early Evidence-based Parent-coaching Interventions for Autism Spectrum Disorder?: A Randomized Controlled Trial
Brief Title: Mindfulness Training and Parent-coaching Interventions for Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Amy Weitlauf, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBSR and P-ESDM; R40MC30769 (Other Grant/Funding Number: Health Resources and Services Administration)
Record Dates: First submitted 2019-03-20; First posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Autism Spectrum Disorder; Parents; Stress
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child-focused Treatment (Active Comparator): Participants in this group participate in 12 sessions of the Parent-implemented Early Start Denver Model (P-ESDM).
  Interventions: Behavioral: Parent-implemented Early Start Denver Model
- Child- and Parent-focused Treatment (Experimental): Participants in this group participate in 12 sessions of the Parent-implemented Early Start Denver Model (P-ESDM). Parents also participate in 6 separate, individual sessions of Mindfulness Based Stress Reduction (MBSR).
  Interventions: Behavioral: Parent-implemented Early Start Denver Model; Behavioral: Mindfulness Based Stress Reduction

INTERVENTIONS:
Behavioral: Parent-implemented Early Start Denver Model — The Parent-implemented Early Start Denver Model (P-ESDM; Rogers et al., 2012) consists of 12 consecutive sessions, each session approximately 1 hour long, that promote parental ability to support and interact with their young children with autism spectrum disorder (ASD). Intervention sessions are conducted in the clinic setting by therapists trained to fidelity by ESDM-certified parent trainers. The manualized intervention has a detailed parent-training curriculum, a specific coaching intervention method, and a therapist fidelity measure. Therapists introduce skills through descriptions, interaction, modeling, coaching, and feedback.
Behavioral: Mindfulness Based Stress Reduction — The Mindfulness Based Stress Reduction (MBSR) protocol is derived from the work by Dykens et al. (2014), which is based on the stress reduction and relaxation program (Kabat-Zinn, 1982, 1990). In this study, it is offered as 6 weekly sessions that run concurrent with the P-ESDM intervention. Participants work one-on-one with a therapist for instruction and practice in mindfulness skills as well as discussions of stress, coping, and homework assignments.
  Arms: Child- and Parent-focused Treatment

SUMMARY:
Caregivers of children with autism spectrum disorder (ASD) report higher levels of depression and distress than caregivers of typically developing children as well as children with other developmental disabilities. The proposed work tests a novel treatment paradigm that blends Mindfulness Based Stress Reduction (MBSR) with an empirically supported and manualized parent training program (Parent-Implemented Early Start Denver Model [P-ESDM]). We hypothesize that directly treating parental distress, while simultaneously providing evidence-based parent training, may greatly enhance child-focused intervention and provide benefits that resonate across the family.

ELIGIBILITY:
Inclusion Criteria:

* Child has diagnosis of autism spectrum disorder
* Child at least 12 months of age but less than 36 months at time of consent
* Parent speaks and reads fluent English

Exclusion Criteria:

* Severe child sensorimotor impairment that would impact participation in treatment

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2018-03-23 (Actual)

PRIMARY OUTCOMES:
Change in parental stress | Baseline to end of study (Every 6 weeks for 9 months)
  The Parenting Stress Index - Short Form, Third Edition (PSI-SF; Abidin, 1995), is a 36-item measure that yields three subscale scores (Parent Child Dysfunctional Interaction, Parenting Distress, Difficult Child) used in present analyses. Each item is rated as by parents as: SA (strongly agree), A (agree), NS (not sure), D (disagree), SD (strongly disagree). Scores are converted to percentile ranks, with higher scores indicating higher levels of stress. Percentile ranks of 15-80 considered typical, and ranks of 81 and above are considered high.
Change in parental depression | Baseline to end of study (Every 6 weeks for 9 months)
  Parents completed the Beck Depression Inventory (BDI; Beck et al., 1984). This instrument consists of 21 items, with higher scores reflecting higher levels of symptomatology.
Change in parental anxiety | Baseline to end of study (Every 6 weeks for 9 months)
  Parents completed the Beck Anxiety Inventory (BAI; Beck et al., 1988). This instrument consists of 21 items, with higher scores reflecting higher levels of symptomatology.
Change in parental mindfulness | Baseline to end of study (Every 6 weeks for 9 months)
  . Parents completed the Five Facet Mindfulness Questionnaire (FFMQ; Baer et al., 2006). The FFMQ consists of 44 items that yield five subscales: Observing, Describing, Acting with Awareness, Nonreactivity, and Nonjudging. Higher scores indicate more mindfulness.
Change in parent relationship quality | Baseline to end of study (Every 6 weeks for 9 months)
  The Dyadic Adjustment Scale (DAS; Spanier, 1989) is a 32-item measure that assesses relationship satisfaction. It includes four subscales scored using a mix of Likert and dichotomous responses. Higher scores indicate higher relationship satisfaction.
Change in parental life satisfaction | Baseline to end of study (Every 6 weeks for 9 months)
  Parents completed the Satisfaction with Life Scale (SLS; Diener et al., 1984). The SLS is a 5-item measure of subjective wellbeing, with each item scored along a 7-point Likert scale (higher scores indicate more satisfaction).
Change in parental sleep quality | Baseline to end of study (Every 6 weeks for 9 months)
  Parents completed the Insomnia Severity Index (ISI; Bastien et al., 2011). The ISI consists of seven items scored from 0-4, with higher scores reflecting more sleep-related impairment.

SECONDARY OUTCOMES:
Change in child autism symptom severity | Baseline, end of treatment (12 weeks), end of study (9 months)
  The Autism Diagnostic Observation Schedule - Second Edition (ADOS-2; Lord et al., 2012) is a standardized clinical observation system for use with people with developmental ages of 12 months and older. Each child completes one module based upon age and language level. This module yields a Calibrated Severity Scores (CSS; range: 1-10). Higher scores reflect higher levels of autism symptoms.
Change in child cognitive functioning | Baseline, end of treatment (12 weeks), end of study (9 months)
  The Mullen Scales of Early Learning (MSEL; Mullen, 1995) is a standardized developmental test for children up to age five years.57 It provides scores in four domains (Visual Reception, Fine Motor, Receptive Language, Expressive Language; M=50, SD=10) and yields an overall ability index termed the Early Learning Composite (ELC; M=100, SD=15). Higher scores reflect higher levels of abilities relative to same-aged peers.
Change in child adaptive behavior | Baseline, end of treatment (12 weeks), end of study (9 months)
  The Vineland Adaptive Behavior Scales - Second Edition (VABS-II; Sparrow et al., 1985), Interview Form is a semistructured interview. It yields four domain standard scores: Communication, Daily Living Skills, Socialization, and Motor Skills (M = 100, SD = 15) as well as an overall Adaptive Behavior Composite (M = 100, SD = 15). High scores reflect better developed adaptive behavior skills.
Change in child problem behaviors | Baseline, end of treatment (12 weeks), end of study (9 months)
  The Achenbach Child Behavior Checklist (CBCL; Achenbach, 2001) yields Internalizing, Externalizing, and Total Problem composite scores. Scores are reported as T scores, with T scores above 65 reflecting clinical significance.
Change in child communication behaviors | Baseline, end of treatment (12 weeks), end of study (9 months)
  The MacArthur CDI Words and Gestures (Fenson et al., 2006) provides a count of parent-reported phrases understood, vocabulary comprehension and production, and actions and gestures. Higher scores indicate more reported language skills.

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Weitlauf, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing procedures will adhere to guidelines established by the NIH sponsored National Database for Autism Research (NDAR). NDAR is a scalable informatics platform for ASD relevant data. NDAR was developed to share data and facilitate collaboration across the ASD field. We will participate in this system for sharing data in hopes that such sharing will accelerate research progress by allowing re-analysis of data, as well as re-aggregation, integration, and rigorous comparison with other data, tools, and methods. We will submit both descriptive and experimental data (http://ndar.nih.gov/).

REFERENCES:
- [Background] Abidin, R. (1995). Parenting Stress Index, 3rd Edition. Lutz, FL: Psychological Assessment Resources.
- [Background] Achenbach, T. M. (2001). Achenbach Child Behavior Checklist. Burlington, VT: ASEBA.
- [Background] Baer RA, Smith GT, Hopkins J, Krietemeyer J, Toney L. Using self-report assessment methods to explore facets of mindfulness. Assessment. 2006 Mar;13(1):27-45. doi: 10.1177/1073191105283504. PMID 16443717
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] Beck AT, Steer RA., Brown GK . Manual for the Beck Depression Inventory-II. 1996. San Antonio: Psychological Corporation.
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Dykens EM, Fisher MH, Taylor JL, Lambert W, Miodrag N. Reducing distress in mothers of children with autism and other disabilities: a randomized trial. Pediatrics. 2014 Aug;134(2):e454-63. doi: 10.1542/peds.2013-3164. Epub 2014 Jul 21. PMID 25049350
- [Background] Fenson, L., Marchman, V., Thal, D., Dale, P., Reznick, S., & Bates, E. (2006). The MacArthur Communicative Development Inventories: User's guide and technical manual (2nd ed.). Baltimore: Brookes.
- [Background] Kabat-Zinn J. An outpatient program in behavioral medicine for chronic pain patients based on the practice of mindfulness meditation: theoretical considerations and preliminary results. Gen Hosp Psychiatry. 1982 Apr;4(1):33-47. doi: 10.1016/0163-8343(82)90026-3. PMID 7042457
- [Background] Kabat-Zinn, J. (1990). Full Catastrophe Living: Using the Wisdom of your Mind to Face Stress, Pain and Illness. New York: Dell Publishing.
- [Background] Lord, C., Rutter, M., DiLavore, P., Risi, S., Gotham, K., & Bishop, S.L. (2012). Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2): Manual. Los Angeles: Western Psychological Services.
- [Background] Mullen, E. M. (1994). Mullen Scales of Early Learning. Circle Pines, MN: American Guidance Service.
- [Background] Rogers SJ, Estes A, Lord C, Vismara L, Winter J, Fitzpatrick A, Guo M, Dawson G. Effects of a brief Early Start Denver model (ESDM)-based parent intervention on toddlers at risk for autism spectrum disorders: a randomized controlled trial. J Am Acad Child Adolesc Psychiatry. 2012 Oct;51(10):1052-65. doi: 10.1016/j.jaac.2012.08.003. Epub 2012 Aug 28. PMID 23021480
- [Background] Spanier, G.B. (1989). Manual for the Dyadic Adjustment Scale. North Tonowanda, NY: Multi-Health Systems.
- [Background] Sparrow, S. D., Cicchetti, D. V., & Balla, D. A. (2005). Vineland-II Adaptive Behavior Scales: Survey Forms Manual. Circle Pines, MN: AGS Publishing.
- [Derived] Weitlauf AS, Broderick N, Stainbrook JA, Taylor JL, Herrington CG, Nicholson AG, Santulli M, Dykens EM, Juarez AP, Warren ZE. Mindfulness-Based Stress Reduction for Parents Implementing Early Intervention for Autism: An RCT. Pediatrics. 2020 Apr;145(Suppl 1):S81-S92. doi: 10.1542/peds.2019-1895K. PMID 32238534